CLINICAL TRIAL: NCT04681742
Title: Feasibility Testing of Cognitive Strategy Training in Post-Concussive Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Anna Boone, Assistant Professor in the Department of Occupational Therapy, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019802
Record Dates: First submitted 2020-12-16; First posted 2020-12-23 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Brain Concussion; Post-Concussion Syndrome
Keywords: metacognition; occupational therapy
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CO-OP Group (Experimental): 10, 45-60 minute Cognitive Orientation to daily Occupational Performance intervention sessions
  Interventions: Behavioral: CO-OP Group

INTERVENTIONS:
Behavioral: CO-OP Group — CO-OP focuses on learning of a global problem-solving strategy, Goal-Plan-Do-Check (GPDC), within the performance of participant-chosen goals. Use of a broadly applicable strategy and meaningful activity ensures the intervention is salient to the participant and increases likelihood of transfer. Uniquely, therapists applying CO-OP use guided discovery methods, such as asking a series of probing questions, to support participants in analyzing their own performance of a given task and generating potential solutions for improving performance. Participants become equipped with these skills through repetitive application of the GPDC process. First, participants identify a specific goal (Goal). Then, participants consider a detailed plan (Plan) for accomplishing the goal. By carrying out the plan (Do) and critically analyzing the results (Check), participants determine how the plan worked. The intervention focuses on learning GPDC with gradual withdrawal of guided discovery methods.

SUMMARY:
This study will evaluate the practicality (i.e. acceptability to stakeholders; outcome battery feasibility; recruitment, retention, and adherence rates) and the preliminary effect of a cognitive strategy training intervention in adults with post-concussive syndrome.

DETAILED DESCRIPTION:
Up to 90% of known traumatic brain injuries are classified as mild, with many more injuries likely going undetected. While each of these individuals experiences somatic, cognitive, and/or affective symptoms acutely following the injury, an estimated 10-15% will continue to experience these symptoms for months up to a year post-injury. The persistence of symptoms for three months or greater is termed post-concussive syndrome (PCS) and can lead to decreases in academics, job performance, leisure, daily life activities, and routines. Traditionally, rehabilitation is either not provided to these individuals or has a specific focus on alleviating impairments (e.g. sustained attention) instead of mitigating effects on daily life function. Transfer of improvements in said impairments is known to be limited. Cognitive Orientation to daily Occupational Performance (CO-OP), a type of metacognitive strategy training, has known positive effects on activity performance outcomes in acquired brain injury (e.g. subacute and chronic stroke; moderate traumatic brain injury)1-5. CO-OP has yet to be evaluated in a sample of individuals with PCS. In sum, (1) CO-OP is an evidence-based intervention for improving activity performance, and (2) it is reasonable to hypothesize that the positive effects of CO-OP may be applied in PCS to overcome similar cognitive difficulties to improve activity performance.

The central research hypothesis is that a functionally-oriented metacognitive strategy training intervention, CO-OP, will be feasible and have a positive effect on activity performance in individuals with PCS syndrome. A single-group, prospective design with outcomes gathered pre-and post-intervention will be used (n=15) to evaluate the acceptability and feasibility of CO-OP in PCS. We will also be evaluating effect size on outcome measures of activity performance and perceptions of the functional impact of PCS symptoms.

Specific Aim 1: Determine the feasibility of CO-OP in Post-Concussive Syndrome. Hypothesis 1.1: Participants will report positive perceptions of the intervention via scores greater than 3 on the Client-Satisfaction Questionnaire. Hypothesis 1.2: The study will demonstrate acceptable recruitment, retention, and adherence rates. Hypothesis 1.3: The proposed assessment battery will be feasible (average completion time <2 hours).

Specific Aim 2: Explore the preliminary effect of CO-OP in a sample of individuals with PCS on activity performance outcomes. Hypothesis 2.1: The CO-OP group will demonstrate improvements in activity performance outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included if have a physician diagnosis of mTBI or if they meet the following criteria for mild traumatic brain injury established by the American Congress of rehabilitation Medicine including a traumatically induced physiological disruption of brain function, as manifested by at least one of the following: any loss of consciousness, any loss of memory for events immediately before or after the accident, any alteration in mental state at the time of the accident (e.g., feeling dazed, disoriented, or confused), and focal neurologic deficit(s) that may or may not be transient; severity of injury should not exceed a loss of consciousness >30 minutes, at 30 minutes post-injury a Glasgow Coma Scale score more severe than 13-15, or post-traumatic amnesia >24 hours.
* One or more post-concussive symptoms persisting for greater than 4 weeks that is inhibiting performance of one or more daily activities
* Age 18-60 years

Exclusion Criteria:

* Any additional severe neurologic or psychiatric conditions
* severe depressive symptoms per a score of >21 on the Patient Health Questionnaire (PHQ-9)
* inability to read, write, and speak English fluently
* lack of transportation to intervention sessions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire-8 | post-intervention only (10 weeks post-baseline)
  Self-report, 8 item measures of intervention acceptability
recruitment rate | calculated at end of intervention (10 weeks post-baseline)
  number enrolled/numberscreened AND Total # enrolled
retention rate | calculated at end of intervention (10 weeks post-baseline)
  number completing study procedures/number enrolled
adherence rate | calculated at end of intervention (10 weeks post-baseline)
  number of sessions attended/Total number of sessions
assessment battery feasibility | calculated at end of intervention (10 weeks post-baseline)
  Time for completion
assessment battery feasibility | calculated at end of intervention (10 weeks post-baseline)
  Percentage of assessment items complete

SECONDARY OUTCOMES:
Canadian Occupation Performance Measure (COPM) | Change from baseline to post-intervention (10 weeks)
  Self-report measures of perceived performance and satisfaction of occupational performance on a 1 to 10 Likert scale.
Neurobehavioral Symptom Inventory | Change from baseline to post-intervention (10 weeks)
  Self-report measure on the severity and impact of common concussive symptoms using a 0 (none) to 4 (very severe) Likert scale.
Pittsburgh Sleep Quality Index | Change from baseline to post-intervention (10 weeks)
  Self-report measure of quality and patterns of sleep using a four point Likert scale
Henry Ford Hospital Headache Disability Inventory | Change from baseline to post-intervention (10 weeks)
  Self-report questionnaire of functional impact of headache symptoms
College of Optometrists in Vision Quality of Life Outcomes Assessment (COVD-QOL) | Change from baseline to post-intervention (10 weeks)
  Self-report measure of functional impact of visual impairments using a five point Likert scale
Dysexecutive Questionnaire | Change from baseline to post-intervention (10 weeks)
  Self-report measure functional impact of dysexecutive symptoms using five point Likert scale.
NIH Toolbox Cognition Battery | Change from baseline to post-intervention (10 weeks)
  Neuropsychological, computer based tests of attention, executive functioning, episodic memory, working memory, language, and processing speed resulting in normative T-scores (mean=50; SD=10)
Weekly Calendar Planning Assessment | Change from baseline to post-intervention (10 weeks)
  Performance-based measure of executive functioning within a calendar planning activity using accuracy and time to completion scores. Alternate forms available.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Boone, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

REFERENCES:
- [Background] Henshaw E, Polatajko H, McEwen S, Ryan JD, Baum CM. Cognitive approach to improving participation after stroke: two case studies. Am J Occup Ther. 2011 Jan-Feb;65(1):55-63. doi: 10.5014/ajot.2011.09010. PMID 21309372
- [Background] Dawson DR, Binns MA, Hunt A, Lemsky C, Polatajko HJ. Occupation-based strategy training for adults with traumatic brain injury: a pilot study. Arch Phys Med Rehabil. 2013 Oct;94(10):1959-63. doi: 10.1016/j.apmr.2013.05.021. Epub 2013 Jun 22. PMID 23796683
- [Background] Dawson DR, Gaya A, Hunt A, Levine B, Lemsky C, Polatajko HJ. Using the cognitive orientation to occupational performance (CO-OP) with adults with executive dysfunction following traumatic brain injury. Can J Occup Ther. 2009 Apr;76(2):115-27. doi: 10.1177/000841740907600209. PMID 19456090
- [Background] McEwen S, Polatajko H, Baum C, Rios J, Cirone D, Doherty M, Wolf T. Combined Cognitive-Strategy and Task-Specific Training Improve Transfer to Untrained Activities in Subacute Stroke: An Exploratory Randomized Controlled Trial. Neurorehabil Neural Repair. 2015 Jul;29(6):526-36. doi: 10.1177/1545968314558602. Epub 2014 Nov 21. PMID 25416738
- [Background] Polatajko HJ, McEwen SE, Ryan JD, Baum CM. Pilot randomized controlled trial investigating cognitive strategy use to improve goal performance after stroke. Am J Occup Ther. 2012 Jan-Feb;66(1):104-9. doi: 10.5014/ajot.2012.001784. PMID 22389945
- [Background] Bergersen K, Halvorsen JO, Tryti EA, Taylor SI, Olsen A. A systematic literature review of psychotherapeutic treatment of prolonged symptoms after mild traumatic brain injury. Brain Inj. 2017;31(3):279-289. doi: 10.1080/02699052.2016.1255779. Epub 2017 Jan 26. PMID 28125305
- [Background] Lundin A, de Boussard C, Edman G, Borg J. Symptoms and disability until 3 months after mild TBI. Brain Inj. 2006 Jul;20(8):799-806. doi: 10.1080/02699050600744327. PMID 17060147
- [Background] Schmitter-Edgecombe M, Seelye AM. Recovery of content and temporal order memory for performed activities following moderate to severe traumatic brain injury. J Clin Exp Neuropsychol. 2012;34(3):256-68. doi: 10.1080/13803395.2011.633497. Epub 2012 Jan 6. PMID 22220505
- [Background] McCrory P, Meeuwisse WH, Aubry M, Cantu RC, Dvorak J, Echemendia RJ, Engebretsen L, Johnston K, Kutcher JS, Raftery M, Sills A, Benson BW, Davis GA, Ellenbogen R, Guskiewicz KM, Herring SA, Iverson GL, Jordan BD, Kissick J, McCrea M, McIntosh AS, Maddocks D, Makdissi M, Purcell L, Putukian M, Schneider K, Tator CH, Turner M. Consensus statement on concussion in sport: the 4th International Conference on Concussion in Sport, Zurich, November 2012. J Athl Train. 2013 Jul-Aug;48(4):554-75. doi: 10.4085/1062-6050-48.4.05. No abstract available. PMID 23855364
- [Background] Taylor CA, Bell JM, Breiding MJ, Xu L. Traumatic Brain Injury-Related Emergency Department Visits, Hospitalizations, and Deaths - United States, 2007 and 2013. MMWR Surveill Summ. 2017 Mar 17;66(9):1-16. doi: 10.15585/mmwr.ss6609a1. PMID 28301451
- [Background] Jagoda AS, Bazarian JJ, Bruns JJ Jr, Cantrill SV, Gean AD, Howard PK, Ghajar J, Riggio S, Wright DW, Wears RL, Bakshy A, Burgess P, Wald MM, Whitson RR. Clinical policy: neuroimaging and decisionmaking in adult mild traumatic brain injury in the acute setting. J Emerg Nurs. 2009 Apr;35(2):e5-40. doi: 10.1016/j.jen.2008.12.010. PMID 19285163
- [Background] King PR, Donnelly KT, Donnelly JP, Dunnam M, Warner G, Kittleson CJ, Bradshaw CB, Alt M, Meier ST. Psychometric study of the Neurobehavioral Symptom Inventory. J Rehabil Res Dev. 2012;49(6):879-88. doi: 10.1682/jrrd.2011.03.0051. PMID 23299259
- [Background] Carpenter JS, Andrykowski MA. Psychometric evaluation of the Pittsburgh Sleep Quality Index. J Psychosom Res. 1998 Jul;45(1):5-13. doi: 10.1016/s0022-3999(97)00298-5. PMID 9720850
- [Background] Jacobson GP, Ramadan NM, Aggarwal SK, Newman CW. The Henry Ford Hospital Headache Disability Inventory (HDI). Neurology. 1994 May;44(5):837-42. doi: 10.1212/wnl.44.5.837. PMID 8190284
- [Background] Carlozzi NE, Tulsky DS, Wolf TJ, Goodnight S, Heaton RK, Casaletto KB, Wong AWK, Baum CM, Gershon RC, Heinemann AW. Construct validity of the NIH Toolbox Cognition Battery in individuals with stroke. Rehabil Psychol. 2017 Nov;62(4):443-454. doi: 10.1037/rep0000195. PMID 29265865
- [Background] Weiner NW, Toglia J, Berg C. Weekly Calendar Planning Activity (WCPA): a performance-based assessment of executive function piloted with at-risk adolescents. Am J Occup Ther. 2012 Nov-Dec;66(6):699-708. doi: 10.5014/ajot.2012.004754. PMID 23106990
- [Background] Bennett PC, Ong B, Ponsford J. Measuring executive dysfunction in an acute rehabilitation setting: using the dysexecutive questionnaire (DEX). J Int Neuropsychol Soc. 2005 Jul;11(4):376-85. doi: 10.1017/s1355617705050423. PMID 16209417
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Maples WC, Hoenes R. The College of Optometrists in Vision Development checklist related to vision function: expert opinions. Optometry. 2009 Dec;80(12):688-94. doi: 10.1016/j.optm.2009.06.003. PMID 19932442
- [Background] Law M, Baptiste S, McColl M, Opzoomer A, Polatajko H, Pollock N. The Canadian occupational performance measure: an outcome measure for occupational therapy. Can J Occup Ther. 1990 Apr;57(2):82-7. doi: 10.1177/000841749005700207. PMID 10104738
- [Background] Ferreira IS, Pinto CB, Saleh Velez FG, Leffa DT, Vulcano de Toledo Piza P, Fregni F. Recruitment challenges in stroke neurorecovery clinical trials. Contemp Clin Trials Commun. 2019 Jul 5;15:100404. doi: 10.1016/j.conctc.2019.100404. eCollection 2019 Sep. PMID 31360793
- [Background] French B, Leathley M, Sutton C, McAdam J, Thomas L, Forster A, Langhorne P, Price C, Walker A, Watkins C. A systematic review of repetitive functional task practice with modelling of resource use, costs and effectiveness. Health Technol Assess. 2008 Jul;12(30):iii, ix-x, 1-117. doi: 10.3310/hta12300. PMID 18547501
- [Background] Waljas M, Iverson GL, Lange RT, Hakulinen U, Dastidar P, Huhtala H, Liimatainen S, Hartikainen K, Ohman J. A prospective biopsychosocial study of the persistent post-concussion symptoms following mild traumatic brain injury. J Neurotrauma. 2015 Apr 15;32(8):534-47. doi: 10.1089/neu.2014.3339. Epub 2015 Feb 25. PMID 25363626